CLINICAL TRIAL: NCT07334184
Title: Role of Magnetic Resonance Imaging in the Diagnostic Evaluation of Adnexal Cystic Lesions.
Brief Title: Role of Magnetic Resonance Imaging in Diagnosis of Adnexal Cystic Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mira Noshey Mehawed, resident, Sohag University
Other Study IDs: Adnexal-Lesions-Radiology-2025
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Adnexal Lesion
Keywords: adnexal lesions
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adnexal cystic lesions cohort: This group consists of female patients of all ages presenting to the Radiology Department at Sohag University Hospital with adnexal cystic lesions detected on ultrasound. Eligible participants have indeterminate or suspicious ultrasound findings and will undergo MRI for further characterization. MRI findings will be correlated with histopathology, surgical data, laboratory results, or follow-up imaging when surgery is not performed.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Magnetic resonance imaging (MRI) of the pelvis will be performed using 1.5T or 3T scanners with a phased-array pelvic coil. The protocol will include axial, sagittal, and coronal T2-weighted images, axial T1-weighted and fat-suppressed T1-weighted images, diffusion-weighted imaging with ADC maps, and dynamic contrast-enhanced sequences when clinically indicated and not contraindicated.

SUMMARY:
This prospective study aims to evaluate the diagnostic accuracy of magnetic resonance imaging (MRI) in characterizing adnexal cystic lesions and differentiating benign from malignant lesions. MRI findings will be correlated with histopathology, surgical data, laboratory results, or follow-up imaging when surgery is not performed, to improve diagnostic confidence and guide appropriate patient management.

DETAILED DESCRIPTION:
Adnexal cystic lesions are commonly encountered in gynecologic imaging and may represent a spectrum of benign and malignant conditions. While ultrasound is the first-line imaging modality due to its accessibility and safety, many adnexal masses remain indeterminate.

Magnetic resonance imaging (MRI) provides superior soft-tissue contrast and multiparametric imaging, including T1-, T2-weighted sequences, diffusion-weighted imaging (DWI), and dynamic contrast-enhanced imaging (DCE), allowing better characterization of adnexal lesions. Features such as solid tissue, papillary projections, thick septa, and restricted diffusion help differentiate malignant from benign lesions.

This prospective study at Sohag University Hospital will include 50 female patients with adnexal cystic lesions detected on ultrasound. MRI findings will be correlated with histopathology, surgical data, laboratory results (CA-125), or follow-up imaging when surgery is not performed. The study aims to assess the diagnostic accuracy of MRI in differentiating benign from malignant adnexal lesions and to improve clinical decision-making regarding patient management.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of any age with adnexal cystic lesions detected by ultrasound
* Adnexal lesions that are indeterminate or suspicious on ultrasound
* Patients who provide written and oral informed consent

Exclusion Criteria:

* Patients unwilling to participate or complete the study
* Contraindications to MRI, including claustrophobia, metallic implants, pacemaker, or prosthetic heart valves

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only biologically female patients with adnexal cystic lesions are eligible, regardless of gender identity.
Study Population: The study population will consist of 50 female patients of all ages presenting to the Radiology Department at Sohag University Hospital with adnexal cystic lesions detected on ultrasound. Eligible participants are those with indeterminate or suspicious ultrasound findings requiring further characterization with MRI. Patients will provide written and oral informed consent prior to inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-26 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of MRI in characterization of adnexal cystic lesions | From MRI examination until final diagnosis (surgery, histopathology, or follow-up imaging), up to 6 months
  Assessment of the diagnostic performance of magnetic resonance imaging (MRI) in differentiating benign from malignant adnexal cystic lesions, using histopathology, intraoperative findings, or follow-up imaging as the reference standard. Diagnostic accuracy will be expressed in terms of sensitivity, specificity, and predictive values.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. All patient data will remain confidential and used solely for the purposes of this study.